CLINICAL TRIAL: NCT05345756
Title: Intraoral Maxillary Protraction Technique With ALT-RAMEC ( Alternate Rapid Maxillary Expansion and Constriction) Protocol Versus Facemask With Maxillary Expansion in Treating Class III Growing Patients With Maxillary Deficiency: A Randomized Clinical Trial
Brief Title: Intraoral Maxillary Protraction Technique vs Facemask Using Alt-RAMEC Protocol for Treatment Class III Growing Patients
Acronym: ALT-RAMEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Andrew Wafdy Nan Demian, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASR1
Record Dates: First submitted 2022-03-26; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral Protraction Technique (Experimental): using intraoral appliance composed of modified lingual arch and miniscrews for indirect anchorage for maxillary protraction after Alt-RAMEC protocol using hybrid expander
  Interventions: Device: Intraoral protraction device
- Extraoral Protraction Technique (Active Comparator): using facemask for maxillary protraction after ALT-RAMEC protocol
  Interventions: Device: Extraoral protraction device

INTERVENTIONS:
Device: Intraoral protraction device — Use of modified lingual arch with indirect anchorage from screws between lower lateral incisor and lower canine to protract maxilla after ALT-RAMEC protocol
  Arms: Intraoral Protraction Technique
Device: Extraoral protraction device — Facemask which is an extraoral appliance used for maxillary protraction
  Arms: Extraoral Protraction Technique

SUMMARY:
The study compares use of intraoral technique for maxillary advancement and extra oral technique with hep of protocol called Alt-RAMEC which depends on repeated expansion and constriction of maxilla to help in maxillary protraction

DETAILED DESCRIPTION:
Delivering hybrid expander supported by 2 miniscrews in palate to perform Alt-RAMEC protocol for 9 weeks then intervention group will start protraction using class iii elastics on modified lingual arch with hooks in canine area and 2 miniscrews labially between lower lateral and canine while control group use face mask for protraction of maxilla

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Growing Patient ( CVM2-CVM3 )
* Skeletal class III (ANB ≤ 0 , A-NV≤ -2 and wits appraisal < -0.3mm)
* Erupted upper and lower first permanent molars and permanent incisors
* Reverse overjet up to -4 mm

Exclusion Criteria:

* History of previous orthodontic treatment
* Cleft lip/palate patients
* Patients with habits that are detrimental to dental occlusion (thumb sucking, tongue thrusting).
* Patients with syndromes

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Maxillary skeletal changes | 8 months
  using lateral cephalometric x-ray to measure maxillary skeletal changes using angular measurements in degrees (SNA)

SECONDARY OUTCOMES:
Mandibular skeletal changes | 8 months
  using lateral cephalometric x-ray to measure mandibular skeletal changes using angular measurements in degrees (SNB)
Maxillary and Mandibular dental changes | 8 months
  using lateral cephalometric x-ray to measure changes using angular measurements in degrees (U1/Palatal plane ,L1/Mandibular plane)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Demian, BDS, Principal Investigator — Cairo University
Locations (1):
- Faculty of Oral and dental medicine - Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No